CLINICAL TRIAL: NCT00656903
Title: High Speed Indocyanine Green Angiography Findings in Induction/PRN Regimen of Intravitreal Ranibizumab Injection for Neovascular Age-Related Macular Degeneration
Brief Title: High Speed Indocyanine Green Angiography Findings in Ranibizumab Treatment for Wet Age-related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080103; 08-EI-0103
Record Dates: First submitted 2008-04-10; First posted 2008-04-11 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2014-08-19

CONDITIONS: Macular Degeneration
Keywords: Lucentis; Indocyanine Green Angiography; Choroidal Neovascularization; Macular Degeneration; Ranibizumab; Age-Related Macular Degeneration; AMD
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will use an eye imaging test called high speed indocyanine green angiography (HS-ICG), which examines leaky vessels in the eye, to try to find out why individuals respond differently to ranibizumab (Lucentis) treatment for wet age-related macular degeneration (AMD). The drug was recently approved by the Food and Drug Administration to treat this disease, but the response to the treatment varies markedly among individuals.

People 50 years of age and older with wet AMD and vision that meets the research protocol criteria may be eligible for this study. Participants undergo the following procedures:

Ranibizumab injections in the study eye once a month for 4 months. Additional injections are given only if the study eye shows signs of bleeding or leaking fluid. The eye is numbed before the injection and the eye area is cleaned with an antiseptic. Antibiotic drops are used for 3 days following the injection to prevent infection.

Clinic visits once a month for 2 years for evaluations to monitor the response to treatment. The evaluations may include the following examinations and tests:

* Eye examination with dilation, optical coherence tomography and photography: The examination measures visual acuity, thickness of your retina (the back of the eye) andeye pressure. Bright lights will also be used so that the doctor can see the back of your eye. Photographs of the eye may be taken.
* Fluorescein angiography to examine the blood vessels in the eye: A dye called fluorescein is injected into a vein in the arm. The dye travels through the veins to the blood vessels in the eyes. A camera takes pictures of the dye as it flows through the blood vessels. This test is done eight times during the study.
* Indocyanine green angiography to examine the blood vessels in the eye: The procedure is the same as for fluorescein angiography, but it uses a dye called indocyanine green. This test is done once a month for the first year of the study and then every 3 months.

DETAILED DESCRIPTION:
Neovascular age-related macular degeneration (AMD) is the leading cause of blindness among elderly in the United States.1 Ranibizumab, an inhibitor of all forms of vascular endothelial growth factor (VEGF), is the first FDA-approved treatment for AMD that significantly improves vision in a quarter to a third of patients and maintains or improves vision in greater than 90% of patients. Ranibizumab decreases the vasopermeability as measured by decreased leakage and fluid on fluorescein (FA) and optical coherence tomography. However, the effect of ranibizumab on the structure and hemodynamics of the choroidal neovascularization (CNV) in AMD, as measured with high-speed indocyanine green angiography (HS-ICG), is not known. The effect or lack of effect on the physical structure of the CNV may help explain the variability of injection frequencies and visual responses among different patients. Since anti-VEGF therapy is designed to inhibit exudative CNV, it is clinically important to develop a standard reproducible method to assess HS-ICG.

In this observational study, our primary objective is to assess whether induction/pro re nata (Induction/PRN) 0.5 mg intravitreal ranibizumab-based treatment for neovascular AMD decreases the size and pattern of the CNV as measured on HS-ICG, as opposed to simply decreasing leakage and fluid as seen on FA and OCT. Although combination therapy is likely the standard treatment for AMD in the future, participants will not be allowed to receive other AMD experimental agents (e.g., immunosuppressive drugs) for either the study or fellow eye while on this study. In consultation with various reading centers, we will attempt to develop a reproducible schema for evaluation of HS-ICG by reviewing pre-treatment and post-treatment HS-ICGs. The grading system development is a secondary objective to achieve a better understanding of anatomical and functional results and an important task for future research. In this study, the first 10 cases will be used to attempt to develop a reproducible grading system. The NEI retina group will review these ICGs and attempt to identify gradable aspects of the lesions that are consistently present on the ICGs. During this time we will continue to collect additional cases for evaluation. The grading system proposed from the first 10 cases will be implemented in the next 10 cases. There will be two independent gradings for each ICG. The results of this dual grading will then be reviewed and problematic areas of grading will be identified. The grading system will be modified based on this experience and reproducibility of the modified grading system will be assessed by re-grading the images in a masked fashion. The modified grading system will be utilized in the next 10 cases. This iterative process will be continued until we have either developed a reproducible and useful grading system or completed the full participant analysis. Another important secondary objective is to examine whether an increased dose of 1 mg of intravitreal ranibizumab-based treatment (administered as 1 mg monthly or 0.5 mg bi-monthly) will decrease leakage and fluid as seen on FA and OCT and/or decrease the size and pattern of CNV on HS-ICG for participants not becoming fluid-free on the standard dose.

ELIGIBILITY:
* INCLUSION CRITERIA:
* The participant must understand and sign the IRB-approved informed consent document for the study.
* The participant must be greater than or equal to 50 years old.
* The participant must be diagnosed with AMD in at least one eye defined by the presence of drusen at least 63 (alpha)m in size.
* The participant must have CNV or associated exudation secondary to AMD as determined by the investigator.
* The participant must have visual acuity of better than 20/400 in the affected eye as measured on an ETDRS chart.
* The participant has retinal photographs and angiography of sufficient quality, allowing assessment of the macular area according to standard clinical practice.
* Women participants of childbearing potential must not be pregnant or breast-feeding, must have a negative pregnancy test at screening, must be willing to undergo a urine pregnancy test throughout the study and must practice an adequate method of birth control. Acceptable methods of birth control include hormonal contraception (birth control pills, injected hormones or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom and spermicide) or surgical sterilization (hysterectomy or tubal ligation).

The participant must be willing and able to comply with the protocol.

EXCLUSION CRITERIA:

* The participant has CNV, associated with other ocular diseases such as pathologic myopia, ocular histoplasmosis or posterior uveitis, etc.
* The participant has geographic atrophy or fibrosis under the fovea that prevents visual acuity improvement at the discretion of the investigator.
* The participant has decreased vision due to retinal disease not attributable to CNV, such as nonexudative forms of AMD, geographic atrophy, inherited retinal dystrophy, uveitis, or epiretinal membrane.
* The participant has any additional ocular diseases that have irreversibly compromised or could likely compromise the visual acuity of the study eye including amblyopia, anterior ischemic optic neuropathy, clinically significant diabetic macular edema, severe non proliferative diabetic retinopathy, or proliferative diabetic retinopathy.
* The participant has decreased vision due to significant media opacity such as corneal disease or cataract, or opacity precluding photography of the retina; a tear of the RPE; a vitelliform-like lesion of the outer retina (e.g., as in pattern dystrophies or basal laminar cuticular drusen), idiopathic parafoveal telangiectasis, or central serous chorioretinopathy.
* The participant has a history of treatment for CNV in the study eye with focal laser photocoagulation (subfoveal, juxtafoveal or extrafoveal), verteporfin/photodynamic therapy, transpupillary thermotherapy, external beam radiation therapy, or other local treatment (such as submacular surgery) that has resulted in significant subfoveal atrophy or fibrosis as determined by the investigator.
* The participant has had previous ranibizumab, bevacizumab or pegaptanib sodium treatments in the study eye less than four weeks prior to enrollment.
* The participant has had prior verteporfin/photodynamic therapy in the fellow eye less than one week prior to enrollment.
* The participant has evidence of ocular toxoplasmosis; external ocular infection, including conjunctivitis; chalazion; significant blepharitis; or aphakia in the study eye.
* The participant has a history of systemic anti-VEGF therapy less than four weeks prior to enrollment.
* The participant has had intraocular surgery (including lens replacement surgery) within six weeks prior to enrollment.
* The participant has a history of (within the last six months), or current ocular or periocular infection (including any history of ocular herpes zoster or simplex).
* The participant has had a prior vitrectomy in the study eye.
* The participant has medical problems that make consistent follow-up over the treatment period unlikely (e.g., stroke, severe MI, end stage malignancy), any contraindications to performing the necessary diagnostic studies (i.e., known allergy to indocyanine green or fluorescein dyes, etc.), or in general is a poor medical risk because of other systemic diseases or active uncontrolled infections.
* The participant has had insertion of a sclera buckle in the study eye.
* The participant has clinical evidence of scleral thinning (defined as an area of blue/grey discoloration of the sclera representing visualization of underlying choroidal tissue through a thinned area of sclera) seen at the time of external eye examination.
* The participant exhibits clinical signs of myopic retinopathy, or has a refraction of > spherical equivalent 8.00D in their current prescription. Pseudophakic participants may be enrolled in this study if there is no funduscopic evidence of degenerative myopia present and if there is no medical history prior to the participants cataract surgery of either myopic retinopathy or a refraction of > spherical equivalent 8.00D.
* The participant has a history of a corneal transplant.
* The participant has infectious conjunctivitis, keratitis, scleritis, or endophthalmitis.
* The participant is currently undergoing treatment for active ocular infection.
* The participant has a shellfish allergy, iodine allergy or liver disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-04-07; Study Completion 2014-08-19

PRIMARY OUTCOMES:
To develop a grading system that can be used to assess the effects of (Induction/PRN) ranibizumab therapy on reducing the neovascular membrane associated with AMD as seen on HS-ICG

SECONDARY OUTCOMES:
Changes in vision; lesion size measured with HS-ICG and FA; leakage measured with FA; changes in retinal thickening measured with OCT; and the safety and tolerability of ranibizumab

CONTACTS AND LOCATIONS:
Overall Officials: Henry E Wiley, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bressler NM, Bressler SB, Fine SL. Age-related macular degeneration. Surv Ophthalmol. 1988 May-Jun;32(6):375-413. doi: 10.1016/0039-6257(88)90052-5. PMID 2457955
- [Background] Laser photocoagulation of subfoveal neovascular lesions in age-related macular degeneration. Results of a randomized clinical trial. Macular Photocoagulation Study Group. Arch Ophthalmol. 1991 Sep;109(9):1220-31. doi: 10.1001/archopht.1991.01080090044025. PMID 1718250
- [Background] Pieramici DJ, Avery RL. Ranibizumab: treatment in patients with neovascular age-related macular degeneration. Expert Opin Biol Ther. 2006 Nov;6(11):1237-45. doi: 10.1517/14712598.6.11.1237. PMID 17049020